CLINICAL TRIAL: NCT01292486
Title: Evaluation of the Spectra Optia® Apheresis System Mononuclear Cell (MNC) Collection Procedure in Multiple Myeloma Patients
Brief Title: Evaluation of the Spectra Optia® Mononuclear Cell Collection Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BCT10-02
Record Dates: First submitted 2011-02-02; First posted 2011-02-09 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with multiple myeloma (Experimental): Multiple myeloma patients who receive autologous stem-cell transplants, collected using the Spectra Optia Apheresis System, following myeloablative therapy. The study is limited to subjects who are expected demonstrate normal neutrophil recovery.
  Interventions: Device: Spectra Optia Apheresis System

INTERVENTIONS:
Device: Spectra Optia Apheresis System — In this study, the safety and effectiveness of the new device will be assessed in two ways. First, MNC collections in growth-factor mobilized cancer patients will be evaluated to confirm that the Spectra Optia is able to collect stem cells. Second, following stem-cell collection and transplant, the number of days required for the collected hematopoetic stem cells to engraft/recover will be compared with historical COBE Spectra engraftment/recovery data.

SUMMARY:
The purpose of this investigation is to establish that hematopoetic stem cells collected on a new centrifugal blood separator, CaridianBCT's Spectra Optia Apheresis System, are able to reconstitute the hematopoetic systems of patients treated with myeloablative therapy, equivalent to hematopoetic cells harvested on the predicate COBE® Spectra platform.

DETAILED DESCRIPTION:
This is a multi-center (3-5) single-arm study that will compare the performance of the Spectra Optia Apheresis System's MNC protocol to that of the historical performance of the COBE Spectra MNC protocol. In order to demonstrate the substantial equivalence of the two devices, a non-inferiority design will be used. The study will enroll patients with multiple myeloma who are to be treated with myeloablative chemotherapy, followed by bone-marrow rescue with an autologous peripheral blood stem-cell transplant. Peripheral blood stem cells will be collected using the Spectra Optia MNC protocol and re-infused following myeloablative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of Multiple Myeloma
* Patients intended to be treated with myeloablative therapy and autologous hematopoetic stem-cell transplant within one month of stem-cell collection
* Patients whose stem-cell mobilization regimen includes G-CSF (granulocyte-colony stimulating factor)
* Males or non-pregnant females, who are 18 years of age or older
* Karnofsky score of ≥70%

Exclusion Criteria:

* Patients with pre-mobilization platelet count < 75,000/µL
* Patients who have received pelvic bone marrow irradiation as part of their conditioning therapy
* Patients who have had a previous hematopoetic stem-cell transplant
* Patients who have had a previous hematopoetic stem-cell collection failure
* Impaired cardiac function, as evidenced by left ventricular ejection fraction <40%.
* Impaired hepatic function, as evidenced by alanine transaminase >2.5 x normal
* Impaired pulmonary function as evidenced by diffusion capacity of the lung for carbon monoxide (adjusted for patient hematocrit, if indicated) or forced expiratory volume in 1 second <50% of predicted
* Impaired renal function, as evidenced by a creatinine clearance < 40 mL/min
* Impaired coagulation, as evidenced by a prothrombin time (PT) > twice normal
* Pregnancy or lactation
* Seropositivity for Human Immunodeficiency Virus-1/2, Hepatitis B Virus, or Hepatitis C Virus
* Documented bacterial or fungal infection that requires intravenous antibiotics to be started or continued while undergoing apheresis collection on the Spectra Optia device
* Subjects enrolled in study protocols that could affect number of CD34+ cells (pluripoten hematopoetic stem stells) collected or kinetics of neutrophil recovery
* Altered mental status, as evidenced by the inability to provide effective informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Bill, MD, Study Director — Terumo BCT
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients requiring a first peripheral blood stem cell collection and transplant for multiple myeloma were recruited at four clinical centers from March through October, 2011.
Pre-assignment Details: This was a single arm study, which evaluated Multiple Myeloma patients who received autologous stem-cell transplants collected using the Spectra Optia Apheresis System, following myeloablative therapy. The study was limited to subjects who were expected to demonstrate normal neutrophil recovery.
Groups:
- All Per Protocol Patients: This was a single arm study, which evaluated Multiple Myeloma patients who received autologous stem-cell transplants collected using the Spectra Optia Apheresis System, following myeloablative therapy. The study was limited to subjects who were expected to demonstrate normal neutrophil recovery.
Period: Overall Study
Arm/Group | All Per Protocol Patients
Started | 32
Completed | 26
Not Completed | 6
Not completed — Protocol Violation | 2
Not completed — Did not meet screening criteria | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With Multiple Myeloma: Multiple myeloma patients requiring myeloablative therapy and a first autologous hematopoetic stem cell transplant.
Arm/Group | Patients With Multiple Myeloma
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 12
Age Continuous [Median (Full Range); unit: years] | 63 [39 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Days Until Neutrophil Recovery Following Peripheral Blood Stem Cell Transplant Minus the Historical Median Day Until Recovery.
Description: Neutrophil recovery is defined as the day on which the peripheral blood absolute neutrophil count exceeds 500/μL (ANC500)for the first of three consecutive measurements obtained on different days following transplant of peripheral blood stem cells in patients treated with myeloablative therapy for their underlying disease.
  As this was a test of non-inferiority, the null hypothesis to be tested (H0) was that the difference between the observed day to neutrophil recovery and the historical median day of neutrophil recovery was greater than two days. At two of the enrolling sites, Duke and Emory Universities, the median day to ANC500 was 12, while at the other two sites, Indiana University and the University of Utah, it was 11 days. Consequently, in the equation below, site specific-historic medians were compared to the observed days to achieve ANC500. H0: D > |2|, where D = Observed median day of neutrophil recovery - Site specific historic median day of neutrophil recovery.
Time Frame: up to 28 days following transplant
Population: Twenty-six patients were evaluable per protocol.
Measure: Median (Full Range); unit: Days
Arm/Group | Patients With Multiple Myeloma
Number analyzed (Participants) | 26
Days | 0 [-1 to 2]
Statistical Analysis 1: Comparison: Patients With Multiple Myeloma; The null hypothesis was that the median day to neutrophil recovery in this study was more than two days longer than historical controls; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 2 days; p < 0.025, Hodges-Lehman estimation; Median Difference (Final Values) = 0, 95% CI 2-sided [0.0 to 0.0]

2. Secondary Outcome: Days Until Platelet Recovery
Description: The time to platelet recovery is defined as the day following stem-cell transplant (Day 0) on which the platelet count exceeds 20,000/μL, for the first of three consecutive measurements obtained on different days, without platelet transfusion support within the preceding 7 days.
Time Frame: up to 28 days following transplant
Population: All per protocol patients for whom platelet recovery data was available.
Measure: Median (Full Range); unit: days
Groups:
- All Per Protocol Patients: Multiple myeloma patients infused with autologous peripheral blood stem cells collected on the Spectra Optia Apheresis System.
Arm/Group | All Per Protocol Patients
Number analyzed (Participants) | 19
days | 20 [11 to 28]

3. Secondary Outcome: CD34+ Cell Collection Efficiency.
Description: Collection efficiency (CE) is defined as the percentage of any given cellular subset, processed by the system, that is collected from the subject.
  CD34+ is a cell surface marker found on pluripotent hematopoeitic stem cells.
Time Frame: up to 7 days
Population: Data to calculate CD34+ cell collection efficiency was available for 39 collections on 24 of 26 per protocol patients.
Measure: Median (Full Range); unit: % of processed CD34+ cells collected
Units Other Than Participants: MNC collections
Arm/Group | All Per Protocol Patients
Number analyzed (Participants) | 24
Number analyzed (MNC collections) | 39
% of processed CD34+ cells collected | 70 [39 to 92]

4. Secondary Outcome: Mononuclear Cel (MNC) Collection Efficiency
Description: Collection efficiency (CE) is defined as the percentage of any given cellular subset, processed by the system, that is collected from the subject.
  Determination of collection efficiency depends on an estimate of the average concentration of target cells in the patient's blood. Because these cells are continuously being removed during the collection, and are undergoing variable replacement from the bone marrow, this estimate will not be completely accurate. Underestimation of the concentration of target cells processed can lead to collection efficiencies of greater than 100%.
Time Frame: up to 7 days
Population: Data was available to calculate MNC collection efficiency on 35 collections performed on 22 of the 26 per protocol patients.
Measure: Median (Full Range); unit: % of processed MNCs that were collected
Units Other Than Participants: MNC collections
Arm/Group | All Per Protocol Patients
Number analyzed (Participants) | 22
Number analyzed (MNC collections) | 35
% of processed MNCs that were collected | 60 [35 to 115]

5. Secondary Outcome: Platelet Collection Efficiency
Description: Platelet contamination of the cell product was measured as the platelet collection efficiency, that is, as the percent of platelets processed that were collected.
Time Frame: up to 7 days
Population: Data to calculate platelet collection efficiency was available for 38 MNC collections on 24 of the 26 per protocol patients.
Measure: Median (Full Range); unit: % of processed platelets collected
Units Other Than Participants: MNC collections
Arm/Group | All Per Protocol Patients
Number analyzed (Participants) | 24
Number analyzed (MNC collections) | 38
% of processed platelets collected | 19 [13 to 38]

6. Secondary Outcome: Hematocrit of MNC Product
Description: The hematocrit of the collected product was used to quantitate Red Blood Cell (RBC) contamination.
Time Frame: 7 days
Population: Data was available from 38 MNC collections from 25 of the 26 per protocol patients.
Measure: Median (Full Range); unit: hematocrit %
Units Other Than Participants: MNC collections
Arm/Group | All Per Protocol Patients
Number analyzed (Participants) | 25
Number analyzed (MNC collections) | 38
hematocrit % | 1.8 [1.1 to 4.5]

7. Secondary Outcome: Granulocyte % of MNC Product
Description: Granulocyte contamination of the MNC product was quantitated as the percent of total product White Blood Cells (WBC) that were segmented granulocytes or bands.
Time Frame: 7 days
Population: Data to calculate the percent of product WBCs that were segmented granulocytes or bands was available for 38 MNC collections on 25 of the 26 per protocol patients.
Measure: Median (Full Range); unit: percentage of product WBCs
Units Other Than Participants: MNC collections
Arm/Group | All Per Protocol Patients
Number analyzed (Participants) | 25
Number analyzed (MNC collections) | 38
percentage of product WBCs | 29.0 [4.0 to 72.0]

ADVERSE EVENTS:
Time Frame: During stem cell collection (3-6 hours) and following reinfusion of collected stem cell product until neutrophil recovery (1-28 days).
Description: Two participants were removed from the study before they underwent a collection on the Spectra Optia Apheresis System and were not at risk.
Arm/Group | Patients With Multiple Myeloma
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Multiple Myeloma (N=30)
Fever and hypotension (Infections and infestations) | 1 (1) — Blood cultures were negative but patient was hospitalized for antibiotic administration. Patient recovered and event judged to unrelated to the device.
Pneumonia/Sepsis (Infections and infestations) | 1 (1) — Required inpatient hospitalization and antibiotics. Patient recovered. Unrelated to the device.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Multiple Myeloma (N=30)
Citrate Reaction (General disorders) | 5 (5)
Fever (Infections and infestations) | 2 (2) — Fever post ahpheresis, pre-apheresis and product cultures negative.Patient recovered.Unrelated to the device. Fever/chills post apheresis, preapheresis blood culture positive.Patient recovered.Unrelated to the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less